CLINICAL TRIAL: NCT02736448
Title: 177Lutethium - Peptide Receptor Radionuclide Therapy (Lu-PRRT) Plus Capecitabine Versus Lu-PRRT in FDG Positive, Gastro-entero-pancreatic Neuroendocrine Tumors: a Randomized Phase II Study.
Brief Title: 177Lutethium - Peptide Receptor Radionuclide Therapy (Lu-PRRT) Plus Capecitabine Versus Lu-PRRT in FDG Positive, Gastro-entero-pancreatic Neuroendocrine Tumors
Acronym: Lu-Ca-S
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Following the publication in the Official Journal of the reclassification of the drug LUTATHERA in band H, it was decided to close the enrolment early on 30/Aug/19.
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.17; 2014-003067-38 (EudraCT Number)
Record Dates: First submitted 2016-04-07; First posted 2016-04-13 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Gastro-entero-pancreatic Neuroendocrine Tumors
Keywords: GEP-NET tumors; Lu-PRRT; 177Lutethium - Peptide Receptor Radionuclide Therapy; gastro-entero-pancreatic neuroendocrine tumors; 18-FDG Positron Emission Tomography (PET) positive; low dose of capecitabine
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm Lu-PRRT-Cap (Experimental): Arm Lu-PRRT-Cap: oral low dose of capecitabine in association with Lu-PRRT (at 3.7 Gbq per cycle x 7 cycles) followed by long acting octreotide or lanreotide (SS-LAR)
  Interventions: Drug: Capecitabine; Drug: Lu-PRRT; Drug: SS-LAR
- Arm Lu-PRRT (Experimental): Arm Lu-PRRT: Lu-PRRT (at 3.7Gbq per cycle x 7 cycles) followed by long acting octreotide or lanreotide (SS-LAR)
  Interventions: Drug: Lu-PRRT; Drug: SS-LAR

INTERVENTIONS:
Drug: Capecitabine — oral low dose of capecitabine
  Arms: Arm Lu-PRRT-Cap
Drug: Lu-PRRT — Lu-PRRT (at 3.7Gbq per cycle x 7 cycles)
Drug: SS-LAR — long acting octreotide or lanreotide

SUMMARY:
This is a randomized phase II, parallel group study. Patients with gastro-entero-pancreatic neuroendocrine tumors (GEP-NET) well differentiated G1 - G2 (ki67≤ 20%) and G3 (ki67≤ 50%), somatostatin receptor (SSR) positive and 18-FDG positive will be enrolled in the study and will be randomly assigned to 2 different arms:

* Arm Lu-PRRT-Cap: oral low dose of capecitabine in association with Lu-PRRT (at 3.7 Gbq per cycle x 7 cycles) followed by long acting octreotide or lanreotide (SS-LAR); OR
* Arm Lu-PRRT: Lu-PRRT (at 3.7 gigabecquerel (Gbq) per cycle x 7 cycles) followed by SS-LAR.

DETAILED DESCRIPTION:
This is a randomized phase II, parallel group study. Patients with gastro-entero-pancreatic neuroendocrine tumors (GEP-NET) well differentiated G1 - G2 (ki67≤ 20%) and G3 (ki67≤ 50%), SSR positive and 18-fluorodeoxyglucose (FDG) positive will be enrolled in the study and will be randomly assigned to 2 different arms:

* Arm Lu-PRRT-Cap: oral low dose of capecitabine in association with Lu-PRRT (at 3.7 Gbq per cycle x 7 cycles) followed by long acting octreotide or lanreotide (SS-LAR); OR
* Arm Lu-PRRT: Lu-PRRT (at 3.7Gbq per cycle x 7 cycles) followed by SS-LAR. The primary objective is to evaluate the progression free survival (PFS) in the two arms.

The secondary objectives are: i) the efficacy (disease control rate, DCR), ii) acute and late toxicity, and iii) overall survival (OS).

The investigators plan to enroll 176 patients during a period of 36 months and a period of 36 months of follow up

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologic diagnosis of gastro-entero-pancreatic neuroendocrine tumor, well differentiated G1 - G2 (ki67≤20%) and G3 (ki67≤50%)
2. Male or Female, aged >18 years
3. Measurable disease according to RECIST 1.1 criteria
4. Patients with documented disease will be admitted to therapeutic phase only if the diagnostic receptor imaging, OctreoScan, with a significant uptake in the tumor (grade 2 or 3, according to Rotterdam scale) and/or PET/CT 68Gallium (68Ga)-peptide images with a tumor uptake at least equal to liver background
5. Patients with documented disease will be admitted to therapeutic phase only if the 18FDG PET/CT is positive with a standardized uptake value (SUV) > 2.5 at least in one documented lesion.
6. Non operable advanced disease
7. Documented progression after standard therapy such as long acting octreotide or lanreotide (SS-LAR), Everolimus in P-NETs or platinum based therapy in G3 patients.
8. Patients have to finish prior standard chemotherapy or therapeutical radiotherapy (less then 25% body surface) at least 6 weeks
9. Life expectancy greater than 6 months.
10. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
11. Adequate haematological, liver and renal function: haemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, total bilirubin ≤ 2.5 X upper normal limit (UNL) , Alanine transaminase (ALT) <2.5 X UNL (< 5 X UNL in presence of liver metastases), creatinine < 2 mg/dL.
12. Concomitant SS-sub-cutaneous assumption is allowed in case of carcinoid syndrome
13. If female of childbearing potential highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials", (2014_09_15 section 4.1) (See Appendix H) are mandatory. Highly effective birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug. Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 6 months after final study drug administration. Two acceptable methods of birth control thus include Condom (barrier method of contraception) and one of the following is required (established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg, bilateral orchiectomy), for more than 6 months.
14. Participant is willing and able to give informed consent for participation in the study.
15. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.

Exclusion Criteria:

1. Ki 67 index > 50%
2. FDG PET negative
3. Patients treated with chemotherapy and therapeutic radiotherapy within 6 weeks
4. More then 25% body surface radiotherapy
5. Patients treated with previous radiometabolic therapy with an adsorbed dose to the kidney more than 23 Gy and 1,2 Gy for the bone marrow or as surrogate of dosimetry, a Total Cumulative Activity (TCA) of >250 millicurie (mCi) of 90Y dotatoc or >800 (mCi) of 177Lutethium (177Lu) dotatate
6. All acute toxic effects of any prior therapy (including surgery radiation therapy, chemotherapy) must have resolved to a grade ≤ 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE)
7. Life expectancy minor than 6 months.
8. ECOG performance status >2
9. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. History of allergic reactions attributed to compounds of similar chemical or biologic composition
12. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
13. Known hypersensitivity to Octreotide and/or Lanreotide, and/or somatostatin correlate peptides
14. Known hypersensitivity to capecitabine or to any of its components
15. Known hypersensitivity to 5 - fluorouracil.
16. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix);

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | up to 72 months
  Progression free survival is defined as the time from the randomization date to the date of first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.

SECONDARY OUTCOMES:
Disease control rate | up to 72 months
  DCR will be evaluated using the new international criteria proposed by the Version 1.1 Response Evaluation Criteria in Solid Tumors (RECIST).
Acute and late toxicity | up to 72 months
  The acute toxicity is the toxicity that occurred within 30 days from the last treatment administration. The late toxicity is the toxicity that occurred over 30 days from the last treatment administration. NCI-CTCAE v. 4.03 will be applied and a profile of adverse events related to the study drug will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Paganelli, MD, Study Chair — IRST IRCCS, Meldola (FC)
Locations (1):
- Irst Irccs, Meldola, FC, Italy

IPD SHARING:
Plan to Share IPD: Undecided